CLINICAL TRIAL: NCT06779019
Title: Breast Enhanced Strategies and Techniques(BEST) (Focus on Chinese Breast Reconstruction) Trial PART 1: Evaluation of Predictive Methods of Reconstruction Outcomes--Flap Perfusion Analysis
Brief Title: a Prospective Study of Surgical Results, Complications and Predictive Values in Chinese Women Breast Reconstruction
Acronym: BEST
Status: Completed | Type: Observational
Sponsor: Peking Union Medical College Hospital (Other)
Collaborators: China Medical Board (CMB) (Unknown)
Responsible Party: Sponsor
Other Study IDs: ZS-3103
Record Dates: First submitted 2025-01-12; First posted 2025-01-16 (Actual); Last update posted 2025-01-16 (Actual); Status verified 2023-10

CONDITIONS: Breast Reconstruction; Flap Necrosis
Keywords: LSCI; ICG; breast reconstruction; implant-based breast reconstruction; flap necrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patients underwent immediate direct-to-implant reconstruction: Patients undergoing nipple-sparing mastectomy (NSM) received flap evaluations for both the nipple-areolar complex (NAC) and the peri-incision skin flap. Perfusion of the skin flap and nipple was assessed using both Laser Speckle Contrast Imaging (LSCI) and Indocyanine Green (ICG) fluorescence imaging at two critical time points: immediately after the mastectomy (prior to immediate reconstruction) and again following reconstruction (after the skin was sutured).
  Interventions: Diagnostic Test: LSCI; Diagnostic Test: ICG (Indocyanine Green)

INTERVENTIONS:
Diagnostic Test: LSCI — LSCI evaluates at 2 timings:immediately after the mastectomy (prior to immediate reconstruction) and again following reconstruction (after the skin was sutured). The perfusion score was calculated by normalizing these values against the perfusion value of a control.
Diagnostic Test: ICG (Indocyanine Green) — Performed immediately after the mastectomy (prior to immediate reconstruction) .Perfusion scores were determined by comparing the fluorescence intensity of the target area to that of the non-surgical region on the contralateral chest wall.

SUMMARY:
This study prospectively evaluates and compares the effectiveness of ICG fluorescence imaging and LSCI in predicting the risk of necrosis following direct-to-implant breast reconstruction.

DETAILED DESCRIPTION:
This study prospectively evaluates and compares the effectiveness of Indocyanine Green (ICG) fluorescence imaging and Laser Speckle Contrast Imaging (LSCI) in predicting the risk of necrosis following direct-to-implant breast reconstruction. The investigation includes both intraoperative and postoperative assessments of flap perfusion, with a focus on identifying specific thresholds for necrosis prediction. By analyzing the sensitivity, specificity, and predictive accuracy of each technique, the study aims to establish their respective strengths and limitations. Additionally, the research aims to explore the feasibility of using these methods in different surgical stages, evaluating their consistency and reliability in monitoring the viability of the skin flap and nipple-areolar complex.

ELIGIBILITY:
Inclusion Criteria:

All patients presenting for implant-base reconstruction immediately after mastectomy

Exclusion Criteria:

delayed reconstruction, expander removal followed by prothesis implant, ICG allergy or intolerance, autologous reconstruction

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: female patients who received mastectomy and immediate direct-to-implant reconstruction
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2024-07-01 (Actual); Study Completion 2024-07-01 (Actual)

PRIMARY OUTCOMES:
necrosis | 3 months
  Signs of necrosis included: (1) swelling or blistering, (2) dark brown or dark blue discoloration of the flap or nipple-areolar complex (NAC), (3) scab formation, (4) wound disruption, and (5) sloughing of the NAC or local flap. Severe necrosis was defined as either (4) or (5), necessitating debridement and secondary closure surgery.

CONTACTS AND LOCATIONS:
Locations (1):
- Pumch, Beijing, Beijing Municipality, China